CLINICAL TRIAL: NCT04211337
Title: A Multicenter, Randomized, Open-label, Phase 3 Trial Comparing Selpercatinib to Physicians Choice of Cabozantinib or Vandetanib in Patients With Progressive, Advanced, Kinase Inhibitor Naïve, RET-Mutant Medullary Thyroid Cancer (LIBRETTO-531)
Brief Title: A Study of Selpercatinib (LY3527723) in Participants With RET-Mutant Medullary Thyroid Cancer
Acronym: LIBRETTO-531
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Loxo Oncology, Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17478; J2G-MC-JZJB (Other: Eli Lilly and Company); 2019-001978-28 (EudraCT Number)
Expanded Access: NCT03906331 (Approved for marketing)
Record Dates: First submitted 2019-12-24; First posted 2019-12-26 (Actual); Results first posted 2024-06-13 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Medullary Thyroid Cancer
Keywords: medullary thyroid carcinoma; targeted therapy
MeSH Terms: conditions — Carcinoma, Medullary | interventions — selpercatinib; cabozantinib; vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Selpercatinib - Treatment A (TRT A) (Experimental): 160 milligrams Selpercatinib administered orally (PO) twice daily (BID).
  Adolescent Dose: 92 milligrams per square meter (mg/m2) BID (not to exceed 160 mg BID).
  Interventions: Drug: Selpercatinib
- Cabozantinib or Vandetanib - Treatment B (TRT B) (Active Comparator): 140 mg Cabozantinib administered orally daily (QD) or 300 mg Vandetanib administered orally QD per physician choice.
  Cabozantinib Adolescent Dose: 40 mg/m2.
  Vandetanib Adolescent Dose:
  * 0.7 - <0.9 - 100 mg every other day (QOD)
  * 0.9 - <1.2 - 100 mg QD
  * 1.2 - <1.6 - 7-day schedule 100 mg - 200 mg - 100 mg - 200 mg - 100 mg - 200 mg - 100 mg
  * ≥1.6 - 200 QD
  Interventions: Drug: Cabozantinib; Drug: Vandetanib

INTERVENTIONS:
Drug: Selpercatinib — Administered orally
  Other Names: LY3527723; LOXO-292
  Arms: Selpercatinib - Treatment A (TRT A)
Drug: Cabozantinib — Administered orally
  Arms: Cabozantinib or Vandetanib - Treatment B (TRT B)
Drug: Vandetanib — Administered orally
  Arms: Cabozantinib or Vandetanib - Treatment B (TRT B)

SUMMARY:
The reason for this study is to see if the study drug selpercatinib is safe and more effective compared to a standard treatment in participants with rearranged during transfection (RET)-mutant medullary thyroid cancer (MTC) that cannot be removed by surgery or has spread to other parts of the body. Participants who are assigned to the standard treatment and discontinue due to progressive disease have the option to potentially crossover to selpercatinib.

DETAILED DESCRIPTION:
Adaptive sample size re-estimation will be performed at interim analysis. The sample size could be increased from approximately 250 to 400 depending on the results of interim analysis.

ELIGIBILITY:
* At least 18 years of age (participants as young as 12 years of age will be allowed if permitted by local regulatory authorities).
* Histologically or cytologically confirmed, unresectable, locally advanced and/or metastatic MTC and no prior history of treatment with kinase inhibitors for advanced/metastatic disease.
* Radiographic progressive disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 at screening compared with a previous image taken within the prior 14 months as assessed by the BICR. Participants with measurable or non-measurable but evaluable disease are eligible; however, participants with non-measurable disease may not have disease limited to bone sites only.
* A defined/acceptable RET gene alteration identified in a tumor, germline deoxyribonucleic acid (DNA) or blood sample.

  * Tumor tissue in sufficient quantity to allow for retrospective central analysis of RET mutation status
* Eastern Cooperative Oncology Group performance status score of 0 to 2.
* Adequate hematologic, hepatic, and renal function and electrolytes.
* Men and women of childbearing potential must agree to use a highly effective contraceptive method during treatment with study drug and for 4 months following the last dose of study drug.
* Ability to swallow capsules.

Exclusion Criteria:

* An additional validated oncogenic driver in MTC if known that could cause resistance to selpercatinib treatment. Examples include, but are not limited to RAS or BRAF gene mutations and NTRK gene fusions.
* Symptomatic central nervous system (CNS) metastases, leptomeningeal carcinomatosis, or untreated spinal cord compression.
* Clinically significant active cardiovascular disease or history of myocardial infarction within 6 months, history of Torsades de pointes, or prolongation of the QTcF >470 milliseconds on more than one electrocardiogram (ECG) during screening. Participants who are intended to receive vandetanib if randomized to the control arm are ineligible if QTcF is >450 milliseconds.
* Active uncontrolled systemic bacterial, viral, or fungal infection or serious ongoing uncontrolled intercurrent illness.
* Active hemorrhage or at significant risk for hemorrhage.
* Other malignancy unless nonmelanoma skin cancer, carcinoma in situ or malignancy diagnosed ≥2 years previously and not currently active. Participants with multiple endocrine neoplasia type 2 (MEN2) associated pheochromocytoma may be eligible.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2026-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM, Study Director — Eli Lilly and Company
Locations (143):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - UCLA Hematology/Oncology - Westwood (Building 100), Los Angeles, California
  - University of California Davis (UC Davis) Comprehensive Cancer Center, Sacramento, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - The James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Hospitals and Clinics, Madison, Wisconsin
- Australia (4):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Perth, Western Australia
- Centre Hospitalier Universitaire de Liège - Domaine Universitaire du Sart Tilman, Liège, Belgium
- Brazil (13):
  - Oncocentro, Belo Horizonte, Minas Gerais
  - Hospital de Cancer de Londrina, Londrina, Paraná
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Centro de Pesquisa Sao Lucas, Campinas, São Paulo
  - Hospital de Clínicas de Ribeirão Preto, Ribeirão Preto, São Paulo
  - Hospital Sírio Libanês, São Paulo, São Paulo
  - Instituto D'Or de Pesquisa e Ensino (IDOR), São Paulo, São Paulo
  - Instituto Nacional de Câncer - INCA, Rio de Janeiro
  - Grupo Oncoclínicas Botafogo, Rio de Janeiro
  - Grupo COI - Clínicas Oncológicas Integradas, Rio de Janeiro
  - Icesp - Instituto Do Câncer Do Estado de São Paulo, São Paulo
  - Centro Paulista de Oncologia Clínica, São Paulo
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- China (19):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Tongren Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital Of Fujian Medical University, Fuzhou, Fujian
  - Gansu Cancer Hospital, Lanzhou, Gansu
  - Sun Yat-Sen University Cancer Centre, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - Jinan Central Hospital, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- Czechia (3):
  - Fakultní nemocnice Brno Bohunice, Brno, Brno-město
  - Fakultni nemocnice Motol, Prague, Praha 5
  - Fakultni nemocnice Olomouc, Olomouc
- France (12):
  - Centre Paul Strauss, Strasbourg, Alsace
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux, Aquitaine
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - Assistance Publique Hôpitaux de Marseille - Hôpital Nord, Marseille, Bouches-du-Rhône
  - Centre François Baclesse, Caen, Calvados
  - Centre Georges François Leclerc, Dijon, Côte-d'Or
  - Institut Claudius Regaud, Toulouse, Haute-Garonne
  - Centre Hospitalier Universitaire d'Angers, Angers, Maine-et-Loire
  - Hopital Claude Huriez - CHU de Lille, Lille, Nord
  - Pitie Salpetriere University Hospital, Paris, Orne
  - Centre Jean Perrin - Centre Régional de Lutte contre le Cancer d'Auvergne, Clermont-Ferrand, Puy-de-Dôme
  - Gustave Roussy, Villejuif, Val-de-Marne
- Germany (8):
  - Klinikum der Universität München Großhadern, München, Bavaria
  - Klinikum der Universität München Großhadern, Würzburg, Bavaria
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsmedizin Johannes Gutenberg Universität Mainz, Mainz, Rhineland-Palatinate
  - Otto-von-Guericke-Universität Magdeburg, Magdeburg, Saxony-Anhalt
  - Charité Universitaetsmedizin Berlin - Campus Mitte, Berlin
  - Hämato-Onkologie Hamburg, Prof. Laack und Partner, Hamburg
- Greece (3):
  - Alexandra Hospital, Athens, Attikí
  - University General Hospital of Heraklion, Heraklion, Irakleío
  - European Interbalkan Medical Center, Thessaloniki, Thessaloniki
- India (6):
  - Regional Cancer Centre - Thiruvananthapuram, Thiruvananthapuram, Kerala
  - HCG Manavata Cancer Centre, Nashik, Maharashtra
  - Grant Medical Foundation - Ruby Hall Clinic, Pune, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - Apollo Gleneagles Hospitals Kolkata, Kolkata, West Bengal
  - Post Graduate Institute of Medical Education & Research (PGIMER), Chandigarh
- Israel (3):
  - Rabin Medical Center, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Hadassah Medical Center, Jerusalem, Jerusalem
- Italy (10):
  - University of Naples Federico II, Napoli, Campania
  - Policlinico Umberto I, Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Istituto Auxologico Italiano, Milan, Milano
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Turin, Piedmont
  - Istituto Nazionale Tumori Regina Elena, Rome, Roma
  - Azienda Ospedaliera Universitaria Pisana, Pisa, Tuscany
  - Ospedale Le Scotte, Siena, Tuscany
  - Istituto Oncologico Veneto IRCCS, Padua, Veneto
  - Azienda Ospedaliera Garibaldi, Catania
- Japan (8):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Osaka University Hospital, Suita, Osaka
  - Japanese Foundation for Cancer Research, Koto, Tokyo
  - National Hospital Organization Kyushu Medical Center, Fukuoka
- Netherlands (4):
  - Maastricht UMC+, Maastricht, Limburg
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek (NKI-AVL), Amsterdam, North Holland
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - University Medical Center Groningen, Groningen
- Poland (2):
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach, Gliwice, Silesian Voivodeship
  - Swietokrzyskie Centrum Onkologii, Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Kielce, Świętokrzyskie Voivodeship
- Russia (6):
  - Clinic Evimed, Chelyabinsk, Chelyabinsk Oblast
  - A. Tsyb Medical Radiological Research Center - branch of the National Medical Research Radiological, Obninsk, Kalužskaja Oblast'
  - Fed State Budgetary Inst "N.N. Blokhin Med Center of Oncology" MHRF, Moscow, Moscow
  - Endocrinology Research Center of Rosmedtechnologies, Moscow, Moscow
  - Saint Petersburg State University, Saint Petersburg, Sankt-Peterburg
  - Saint-Petersburg City Clinical Oncology Dispensary, Saint Petersburg, Sankt-Peterburg
- South Korea (6):
  - Chungbuk National University Hospital, Jungbuk, Chungcheongbuk-do [Chungbuk]
  - National Cancer Center, Goyang-si, Kyǒnggi-do
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
- Spain (12):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Catalunya [Cataluña]
  - Institut Català d'Oncologia (ICO) - Girona, Girona, Girona [Gerona]
  - Clinica Universidad de Navarra, Madrid, Madrid, Comunidad de
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital Universitario La Paz, Madrid, Madrid, Comunidad de
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (6):
  - Velindre Cancer Centre, Cardiff, Cardiff [Caerdydd Gb-crd]
  - Weston Park Hospital, Sheffield, England
  - Gartnavel General Hospital, Glasgow, Glasgow City
  - Royal Marsden Hospital (Chelsea), London, Kensington and Chelsea
  - University College London Hospital, London, London, City of
  - Royal Marsden Hospital (Sutton), London, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Hadoux J, Elisei R, Brose MS, Hoff AO, Robinson BG, Gao M, Jarzab B, Isaev P, Kopeckova K, Wadsley J, Fuhrer D, Keam B, Bardet S, Sherman EJ, Tahara M, Hu MI, Singh R, Lin Y, Soldatenkova V, Wright J, Lin B, Maeda P, Capdevila J, Wirth LJ; LIBRETTO-531 Trial Investigators. Phase 3 Trial of Selpercatinib in Advanced RET-Mutant Medullary Thyroid Cancer. N Engl J Med. 2023 Nov 16;389(20):1851-1861. doi: 10.1056/NEJMoa2309719. Epub 2023 Oct 21. PMID 37870969
- [Derived] Wirth LJ, Brose MS, Elisei R, Capdevila J, Hoff AO, Hu MI, Tahara M, Robinson B, Gao M, Xia M, Maeda P, Sherman E. LIBRETTO-531: a phase III study of selpercatinib in multikinase inhibitor-naive RET-mutant medullary thyroid cancer. Future Oncol. 2022 Sep;18(28):3143-3150. doi: 10.2217/fon-2022-0657. Epub 2022 Aug 15. PMID 35969032
- [Derived] Jaber T, Dadu R, Hu MI. Medullary thyroid carcinoma. Curr Opin Endocrinol Diabetes Obes. 2021 Oct 1;28(5):540-546. doi: 10.1097/MED.0000000000000662. PMID 34292174
- See also: A Study of Selpercatinib (LY3527723) in Participants With RET-Mutant Medullary Thyroid Cancer — https://trials.lillytrialguide.com/en-US/trial/MAk6ymq4v0xp57E7leZ7P

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: If a participant has a recorded death on study, or is alive and being followed but off treatment, then the participant can be considered to be study completer.
  Participants randomized to the Cabozantinib or Vandetanib arm will be allowed to crossover to receive the investigational product at the time of Blinded Independent Committee Review (BICR) confirmed radiographic progression.
Groups:
- Selpercatinib - Treatment A (TRT A): 160 milligrams (mg) Selpercatinib administered orally (PO) twice daily (BID).
  Adolescent Dose: 92 milligrams per square meter (mg/m2) BID (not to exceed 160 mg BID).
Period: Overall Study
Arm/Group | Selpercatinib - Treatment A (TRT A) | Cabozantinib or Vandetanib - Treatment B (TRT B)
Started | 193 | 98
Received at Least One Dose of Study Drug | 193 | 97
Completed | 18 | 56
Not Completed | 175 | 42
Not completed — On Treatment | 175 | 40
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants, even if a participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol.
Groups:
- Selpercatinib (TRT A): 160 milligrams Selpercatinib administered orally (PO) twice daily (BID).
  Adolescent Dose: 92 mg/m2 BID (not to exceed 160 mg BID).
- Cabozantinib or Vandetanib (TRT B): 140 mg Cabozantinib administered orally daily (QD) or 300 mg Vandetanib administered orally QD per physician choice.
  Cabozantinib Adolescent Dose: 40 mg/m2.
  Vandetanib Adolescent Dose:
  * 0.7 - <0.9 - 100 mg every other day (QOD)
  * 0.9 - <1.2 - 100 mg QD
  * 1.2 - <1.6 - 7-day schedule 100 mg - 200 mg - 100 mg - 200 mg - 100 mg - 200 mg - 100 mg
  * ≥1.6 - 200 QD
- Total: Total of all reporting groups
Arm/Group | Selpercatinib (TRT A) | Cabozantinib or Vandetanib (TRT B) | Total
Number analyzed (Participants) | 193 | 98 | 291
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 143 | 72 | 215
  >=65 years | 49 | 26 | 75
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 30 | 108
  Male | 115 | 68 | 183
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 9 | 3 | 12
  Unknown or Not Reported | 181 | 94 | 275
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 43 | 24 | 67
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 116 | 52 | 168
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 29 | 20 | 49
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 4 | 15
  Czechia | 6 | 0 | 6
  Japan | 5 | 1 | 6
  United Kingdom | 9 | 3 | 12
  India | 9 | 2 | 11
  Russia | 15 | 6 | 21
  Spain | 9 | 3 | 12
  Greece | 3 | 1 | 4
  Canada | 1 | 1 | 2
  Netherlands | 6 | 3 | 9
  South Korea | 10 | 2 | 12
  Belgium | 1 | 0 | 1
  China | 14 | 16 | 30
  Taiwan | 4 | 1 | 5
  Brazil | 20 | 13 | 33
  Poland | 15 | 10 | 25
  Italy | 14 | 6 | 20
  Israel | 1 | 0 | 1
  Australia | 9 | 2 | 11
  France | 24 | 18 | 42
  Germany | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) by Blinded Independent Central Review (BICR)
Description: PFS is defined as the time from randomization until the occurrence of documented disease progression by the BICR, per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria, or death from any cause in the absence of BICR-documented progressive disease.
  Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Baseline to Progressive Disease or Death from Any Cause, Whichever Occurs First, Up to 39 Months
Population: All randomized participants, even if a participant did not take the assigned treatment, did not receive the correct treatment, or otherwise did not follow the protocol. Censored participants: Selpercatinib - 167; Cabozantinib or Vandetanib - 66
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Selpercatinib (TRT A) | Cabozantinib or Vandetanib (TRT B)
Number analyzed (Participants) | 193 | 98
Months | NA [NA to NA] — Data unavailable due to high censoring. | 16.76 [12.22 to 25.10]
Statistical Analysis 1: Comparison: Selpercatinib (TRT A) vs Cabozantinib or Vandetanib (TRT B); Test type: Superiority; p < 0.0001, Log Rank; Stratified by RET mutation type (M918T vs. Others) and intended treatment if randomized to Arm B (Vandetanib vs. Cabozantinib); Hazard Ratio (HR) = 0.280, 95% CI 2-sided [0.165 to 0.475] — Stratified by RET mutation type (M918T vs. Others) and intended treatment if randomized to Arm B (Vandetanib vs. Cabozantinib)

2. Secondary Outcome: Treatment Failure-Free Survival (TFFS) by Blinded Independent Committee Review (BICR)
Description: TFFS by BICR is defined as the time from randomization to the first occurrence of:
  * documented radiographic disease progression per RECIST 1.1 as assessed by BICR; or
  * unacceptable toxicity leading to treatment discontinuation as assessed by the investigator.
  Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
  To qualify as an event, the toxicity must be from an intolerable AE (defined as any study drug-related AE that meets protocol guidance for treatment discontinuation, with the exception of alopecia); or death (due to any cause).
Time Frame: Baseline to Progressive Disease, Unacceptable Toxicity or Death from Any Cause Up to 39 Months
Population: All randomized participants, even if a participant did not take the assigned treatment, did not receive the correct treatment, or otherwise did not follow the protocol. Censored participants: Selpercatinib - 166; Cabozantinib or Vandetanib - 61
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Selpercatinib (TRT A) | Cabozantinib or Vandetanib (TRT B)
Number analyzed (Participants) | 193 | 98
Months | NA [NA to NA] — Data not available due to high censoring. | 13.93 [11.27 to 25.10]
Statistical Analysis 1: Comparison: Selpercatinib (TRT A) vs Cabozantinib or Vandetanib (TRT B); Test type: Superiority; p < 0.0001, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.254, 95% CI 2-sided [0.153 to 0.423] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Overall Response Rate (ORR): Percentage of Participants With Complete Response (CR) or Partial Response (PR) by BICR
Description: ORR is defined as the number of participants who achieved the best overall response (BOR) of CR or PR divided by the total number of participants randomized to each treatment arm. ORR per RECIST 1.1 as assessed by BICR.
Time Frame: Baseline through Disease Progression or Death Up to 39 Months
Population: All randomized participants, even if a participant did not take the assigned treatment, did not receive the correct treatment, or otherwise did not follow the protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Selpercatinib (TRT A) | Cabozantinib or Vandetanib (TRT B)
Number analyzed (Participants) | 193 | 98
Percentage of Participants | 69.4 [62.4 to 75.8] | 38.8 [29.1 to 49.2]
Statistical Analysis 1: Comparison: Selpercatinib (TRT A) vs Cabozantinib or Vandetanib (TRT B); Test type: Superiority; p < 0.0001, Clopper-Pearson method — Stratified by RET mutation type (M918T vs. Others) and intended treatment if randomized to Arm B (Vandetanib vs. Cabozantinib); Odds Ratio (OR) = 3.7, 95% CI 2-sided [2.2 to 6.3]

4. Secondary Outcome: Duration of Response (DoR) by BICR
Description: DoR by BICR is defined as the time from the date that measurement criteria for complete response (CR) or partial response (PR) (whichever is first recorded) are first met by the BICR or investigator assessment, as applicable, until the first date that disease is recurrent or documented disease progression is observed, per RECIST 1.1 criteria, or the date of death from any cause in the absence of documented disease progression or recurrence. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Date of CR or PR to Date of Disease Progression or Death Due to Any Cause Up to 39 Months
Population: All randomized participants, even if a participant did not take the assigned treatment, did not receive the correct treatment, or otherwise did not follow the protocol. Censored participants: Selpercatinib - 119, Cabozantinib or Vandetanib - 25
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Selpercatinib (TRT A) | Cabozantinib or Vandetanib (TRT B)
Number analyzed (Participants) | 134 | 38
Months | NA [NA to NA] — Data not available due to high censoring. | 16.56 [10.41 to NA] — Upper level Confidence Interval not available due to high censoring.
Statistical Analysis 1: Comparison: Selpercatinib (TRT A) vs Cabozantinib or Vandetanib (TRT B); Test type: Superiority; p = 0.0004, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.275, 95% CI 2-sided [0.129 to 0.587]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from randomization until death from any cause. If the participant is alive or lost to follow-up at the time of data analysis, OS data will be censored on the last date the participant is known to be alive.
Time Frame: Baseline
Reporting Status: Not Posted, anticipated posting 2027-02

6. Secondary Outcome: PFS2 by Investigator
Description: Progression-free survival 2 (PFS2) is defined as the time from randomization to disease progression (radiographic or symptomatic progression as determined by the investigator) on the next line of treatment or death from any cause in the absence of observed disease progression. If the participant is alive at the cutoff for analysis, and disease progression has not been observed, PFS2 data will be censored on the latest date of last progression-free assessment or start of the next line of treatment.
Time Frame: Baseline
Reporting Status: Not Posted, anticipated posting 2027-02

7. Secondary Outcome: Comparative Tolerability: Number of Weeks With High Side Effect Bother Based Score of 3 or 4 on the Functional Assessment of Cancer Therapy Item GP5 (FACT-GP5)
Description: Comparative tolerability defined as a comparison of the proportion of time on treatment with high side effect bother as assessed by the FACT-GP5. The FACT-GP5 is a single question used to assess the overall bother of the treatment side effects. It is scored using a 5-point rating scale (0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; and 4 = very much), where lower scores reflect less bother from treatment side effects.
  Time with high side effect bother (i.e.) score of 3 or 4 is reported here and was derived as follows: cumulative amount of time, in weeks, during which a participant reports high side effect bother divided by the total duration of therapy (weeks), derived as (date of last study treatment dose - date of first study treatment dose + 1) divided by 7.
Time Frame: Baseline to Progressive Disease, Unacceptable Toxicity or Death from Any Cause Up to 39 Months
Population: All participants who received the first dose of study treatment prior to the interim efficacy analysis and at least 6 months prior to the data cutoff date. Analysis of tolerability will be based on the actual treatment a participant received on the first study treatment administration regardless of which treatment they were randomized to receive ("as treated").
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Selpercatinib (TRT A) | Cabozantinib or Vandetanib (TRT B)
Number analyzed (Participants) | 145 | 77
Weeks | 0.08 (0.169) | 0.24 (0.304)
Statistical Analysis 1: Comparison: Selpercatinib (TRT A) vs Cabozantinib or Vandetanib (TRT B); Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.23 to -0.10]

8. Secondary Outcome: The Concordance of the Local Lab and the Central Lab RET Results: Percentage of Participants With RET-Positive Specimens as Called by the Central Lab, Which is Also RET-Positive as Called by a Local Lab (Positive Percent Agreement)
Time Frame: Baseline
Reporting Status: Not Posted, anticipated posting 2027-02

ADVERSE EVENTS:
Time Frame: Baseline up to 39 months
Description: All randomized participants who received at least 1 dose (including a partial dose) of study treatment. Analysis of safety data will be based on the actual treatment a participant received on the first study treatment administration regardless of which treatment they were randomized to receive ("as treated"). Gender specific events occurring only in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- Cabozantinib or Vandetanib - Treatment B (TRT B): 140 mg Cabozantinib administered orally daily (QD) or 300 mg Vandetanib administered orally QD per physician choice.
  Cabozantinib Adolescent Dose: 40 mg/m2.
  Vandetanib Adolescent Dose:
  0.7 - <0.9 - 100 mg every other day (QOD) 0.9 - <1.2 - 100 mg QD 1.2 - <1.6 - 7-day schedule 100 mg - 200 mg - 100 mg - 200 mg - 100 mg - 200 mg - 100 mg
  ≥1.6 - 200 QD
Arm/Group | Selpercatinib - Treatment A (TRT A) | Cabozantinib or Vandetanib - Treatment B (TRT B)
All-Cause Mortality (participants affected / at risk) | 8/193 | 10/97
Serious Adverse Events (participants affected / at risk) | 43/193 | 27/97
Other Adverse Events (participants affected / at risk) | 184/193 | 96/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Selpercatinib - Treatment A (TRT A) (N=193) | Cabozantinib or Vandetanib - Treatment B (TRT B) (N=97)
Polycythaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (2) | 0 (0)
Adrenocortical insufficiency acute (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 1 (1) | 0 (0)
Anal cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (3)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (5) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (2) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (2) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis escherichia coli (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis viral (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1)
Fibrin d dimer increased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/115 (1) | 0/67 (0)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Motor dysfunction (Nervous system disorders) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1/78 (1) | 0/30 (0)
Pelvic organ prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Colporrhaphy (Surgical and medical procedures) | 1/78 (1) | 0/30 (0)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Proctectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 4 (4)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Selpercatinib - Treatment A (TRT A) (N=193) | Cabozantinib or Vandetanib - Treatment B (TRT B) (N=97)
Anaemia (Blood and lymphatic system disorders) | 11 (12) | 10 (16)
Leukopenia (Blood and lymphatic system disorders) | 10 (13) | 6 (7)
Lymphopenia (Blood and lymphatic system disorders) | 10 (16) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 3 (6) | 8 (17)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (5) | 9 (10)
Hypothyroidism (Endocrine disorders) | 12 (18) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 10 (16) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 19 (28) | 14 (30)
Abdominal pain upper (Gastrointestinal disorders) | 16 (19) | 7 (12)
Ascites (Gastrointestinal disorders) | 11 (11) | 0 (0)
Constipation (Gastrointestinal disorders) | 31 (58) | 12 (14)
Diarrhoea (Gastrointestinal disorders) | 51 (116) | 59 (195)
Dry mouth (Gastrointestinal disorders) | 61 (72) | 10 (12)
Dyspepsia (Gastrointestinal disorders) | 19 (21) | 8 (14)
Dysphagia (Gastrointestinal disorders) | 6 (7) | 6 (7)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 (11) | 8 (11)
Nausea (Gastrointestinal disorders) | 20 (36) | 31 (54)
Oral pain (Gastrointestinal disorders) | 3 (3) | 5 (11)
Stomatitis (Gastrointestinal disorders) | 7 (8) | 15 (32)
Toothache (Gastrointestinal disorders) | 3 (4) | 5 (5)
Vomiting (Gastrointestinal disorders) | 15 (20) | 20 (25)
Asthenia (General disorders) | 21 (31) | 24 (40)
Face oedema (General disorders) | 15 (19) | 2 (3)
Fatigue (General disorders) | 36 (61) | 20 (43)
Mucosal inflammation (General disorders) | 14 (17) | 25 (79)
Oedema peripheral (General disorders) | 32 (42) | 2 (2)
Pain (General disorders) | 7 (8) | 6 (9)
Pyrexia (General disorders) | 22 (29) | 2 (2)
Hepatic cytolysis (Hepatobiliary disorders) | 5 (10) | 5 (7)
Covid-19 (Infections and infestations) | 19 (19) | 17 (17)
Urinary tract infection (Infections and infestations) | 11 (13) | 8 (11)
Alanine aminotransferase increased (Investigations) | 51 (139) | 33 (57)
Aspartate aminotransferase increased (Investigations) | 46 (105) | 37 (60)
Blood alkaline phosphatase increased (Investigations) | 19 (37) | 13 (16)
Blood bilirubin increased (Investigations) | 21 (47) | 8 (12)
Blood creatinine increased (Investigations) | 18 (41) | 2 (4)
Blood lactate dehydrogenase increased (Investigations) | 9 (11) | 14 (17)
Blood thyroid stimulating hormone increased (Investigations) | 13 (16) | 13 (14)
Electrocardiogram qt prolonged (Investigations) | 26 (67) | 13 (22)
Neutrophil count decreased (Investigations) | 10 (24) | 9 (22)
Platelet count decreased (Investigations) | 12 (16) | 7 (17)
Weight decreased (Investigations) | 10 (10) | 27 (49)
Weight increased (Investigations) | 22 (44) | 2 (2)
White blood cell count decreased (Investigations) | 17 (33) | 9 (21)
Decreased appetite (Metabolism and nutrition disorders) | 23 (29) | 27 (45)
Hypercalcaemia (Metabolism and nutrition disorders) | 10 (22) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 13 (21) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 20 (43) | 25 (56)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (16) | 15 (33)
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 (15) | 7 (13)
Hyponatraemia (Metabolism and nutrition disorders) | 10 (24) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (16) | 12 (16)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (18) | 11 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 5 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (19) | 5 (6)
Dizziness (Nervous system disorders) | 11 (13) | 10 (15)
Dysgeusia (Nervous system disorders) | 10 (10) | 16 (19)
Headache (Nervous system disorders) | 44 (70) | 20 (22)
Paraesthesia (Nervous system disorders) | 4 (6) | 7 (7)
Insomnia (Psychiatric disorders) | 6 (10) | 5 (5)
Haematuria (Renal and urinary disorders) | 1 (1) | 8 (13)
Proteinuria (Renal and urinary disorders) | 3 (3) | 23 (44)
Erectile dysfunction (Reproductive system and breast disorders) | 12/115 (15) | 0/67 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (25) | 7 (8)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 5 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (17) | 5 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 6 (8)
Acne (Skin and subcutaneous tissue disorders) | 4 (5) | 6 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (10) | 7 (7)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 13 (16) | 11 (11)
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (10)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 (7) | 41 (93)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (9) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 28 (36) | 20 (39)
Hypertension (Vascular disorders) | 82 (158) | 39 (76)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/37/NCT04211337/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/37/NCT04211337/SAP_001.pdf